CLINICAL TRIAL: NCT00065624
Title: Antioxidant Functions of Lipoic Acid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT001062-01A2 (NIH)
Record Dates: First submitted 2003-07-29; First posted 2003-07-31 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-09

CONDITIONS: Hypercholesterolemia
Keywords: Lipoic acid; F2-isoprostanes; endothelial dysfunction; natural product
MeSH Terms: conditions — Hypercholesterolemia | interventions — Thioctic Acid

INTERVENTIONS:
Drug: lipoic acid

SUMMARY:
The goal of this study is to determine whether a short treatment with lipoic acid, an antioxidant used in the treatment of diabetic neuropathy, improves blood vessel reactivity and decreases oxidant stress in persons with elevated blood cholesterol.

DETAILED DESCRIPTION:
As per Brief Summary

ELIGIBILITY:
Inclusion criteria:

* Lipid criteria for inclusion are a plasma LDL between 160 and 190 mg/dl (total cholesterol usually 240-285 mg/dl)
* Less than 2 coronary risk factors, and already on a cholesterol-lowering diet.

Exclusion criteria:

* Overt or clinical atherosclerosis
* Diabetes
* Currently taking cholesterol-lowering medication.
* Subjects with other lipid disorders
* Subjects taking supplemental lipoic acid, vitamin C, or vitamin E.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2003-11; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M May, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States